CLINICAL TRIAL: NCT05259410
Title: The Safety and Efficacy of Time Restricted Eating Alone or Combined the Mediterranean Diet During Chemotherapy for Breast Cancer
Brief Title: Time Restricted Eating During Chemotherapy for Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Kelsey Nicole Dipman Gabel, Clinical Assistant Professor, Postdoctoral Research Associate, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0974
Record Dates: First submitted 2022-01-26; First posted 2022-02-28 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Time restricted eating (Experimental): Participants will eat all food within the same self selected 8 hour window daily.
  Interventions: Behavioral: TRE
- Standard care (No Intervention): Current standard care is to eat enough calories and protein to maintain weight and lean mass.
- Med TRE (Experimental): Participants will eat a mediterranean style diet within the same self selected 8 hour window daily.
  Interventions: Behavioral: MedTRE

INTERVENTIONS:
Behavioral: TRE — All food eaten within the same self-selected 8 hour eating window daily, water fasting the remaining hours of the day.
  Arms: Time restricted eating
Behavioral: MedTRE — A mediterranean style diet will be eaten within the same self-selected 8 hour eating window daily, water fasting the remaining hours of the day.
  Arms: Med TRE

SUMMARY:
Breast cancer is the most common cancer in the United States however, little is known about how diet can affect cancer treatment. Pre-clinical murine studies report intermittent fasting increases effectiveness of chemotherapy and decreases treatment related adverse events. The proposed research will demonstrate that time restricted eating, a form of intermittent fasting, will improve treatment related outcomes, patient related outcomes, and limit treatment related weight gain and fat mass accretion.Time restricted eating combined with a mediterranean diet will also be feasible and improve cardiometabolic risk more than TRE alone or standard care.

DETAILED DESCRIPTION:
Current standard of care during chemotherapy for breast cancer suggests enough daily calories and protein to maintain body weight and avoid muscle loss. However, this approach may be antiquated given weight gain is common during treatment and emerging pre-clinical and clinical evidence suggest that fasting during chemotherapy may improve clinical and patient-reported outcomes. For example, preliminary human trials examining the fasting mimicking diet (very low-calorie, low-protein diet 1-week per month) or short term fasting (48-120 hours (h)), known as periodic fasting, surrounding chemotherapy may increase effectiveness of treatment and decrease side effects related to chemotherapy. Yet these diets have low adherence, side effects of their own, and may increase patient burden and decrease quality of life. In contrast, time restricted eating (TRE) is a form of intermittent fasting with high adherence that may have similar positive effects on treatment outcomes without the untoward side-effects. Moreover, TRE may have beneficial effects on glucose regulation and body composition (i.e., decreased weight and body fat gain) suggesting the potential importance of this regimen to breast cancer recurrence. TRE is extremely accessible with no calorie counting or financial burden to the patient, individuals just shorten their eating window daily. However TRE also does no address diet quality. The Mediterranean diet has also been shown to improve patient and treatment outcomes in this population. The additive effect might be even more beneficial. Despite the potential benefits, TRE alone or TRE combined with a mediterranean has not been investigated in breast cancer patients during chemotherapy treatment. We aim to test the safety and feasibility of 8-h TRE compared to TRE combined with a mediterranean style diet among female breast cancer patients initiating chemotherapy for stage I-III breast cancer. We further strive to examine the preliminary efficacy of TRE or TRE with the mediterranean diet on treatment related outcomes, treatment related side effects, patient-reported quality of life and fatigue, blood-based metabolic markers and body/weight adiposity compared to the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-99 at time of consent
* ECOG 0 or 1
* Breast cancer to meet histologically confirmed Stage I-III.
* Demonstrates adequate organ function (absolutely neutrophil count ≥ 1,500/μL).
* All screening labs to be obtained within 30 days prior to registration.
* Able to provide written informed consent and HIPAA authorization for release of personal health information, via an approved UIC Institutional Review Board (IRB) informed consent form and HIPAA authorization.
* Women of childbearing potential must not be pregnant or breast-feeding. A negative serum or urine pregnancy test is required per institutional practice guidelines.
* As determined at the discretion of the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

* Women with metastatic disease or type 1 or 2 diabetes
* Women with BMI ≥ 40kg/m2 and < 25kg/m2
* Women who are pregnant. A negative serum or urine pregnancy test is required per institutional practice guidelines.
* Night shift workers
* Women with a history of eating disorders
* Enrolled participants with a significant weight loss or weight gain within 3 months of the study (weight gain or loss >4kg)
* Active infection requiring systemic therapy
* Uncontrolled HIV/AIDS or active viral hepatitis
* Pregnant or nursing
* Any prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of this investigational regimen, as determined by the treating medical oncologist.
* Any mental or medical condition that prevents the patient from giving informed consent or participating in the trial.
* Other major comorbidity, as determined by study PI
* Illicit drug use or excessive use of alcohol (i.e., > 2 drinks/day)
* Currently participating in Weight Watcher's or another weight loss program
* Myocardial infarction
* Stroke
* Congestive heart failure
* Chronic hepatitis
* Cirrhosis
* Chronic pancreatitis
* History of solid organ transplantation

Ages: 25 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility 8-h TRE | 12 weeks
  enrollment rate

SECONDARY OUTCOMES:
Relative dose intensity | 12 weeks
  dose intensity between groups
Treatment side effects | 12 weeks
  Side effects
EROTC quality of life score | 12 weeks
  quality of life will be measured by EORTC questionnaire at week 1, 6, and 12
Body weight change | 12 weeks
  body weight
Body composition | 12 weeks
  body fat percentage
Change in glucose | 12 weeks
  glucose
Change in insulin | 12 weeks
  insulin

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey Gabel, MS, RD, PhD, Principal Investigator — UIC
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No